CLINICAL TRIAL: NCT02808754
Title: Remote Ischemic Preconditioning for Carotid Endarterectomy
Acronym: RIP-CEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Natalie Domenick Sridharan, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO16030479; UL1TR001857 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Carotid Stenosis; Endarterectomy, Carotid
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients in the usual care arm will undergo CEA without RIPC.
- Remote Ischemic Preconditioning (Experimental): Patients in the RIPC arm will undergo CEA with RIPC.
  Interventions: Procedure: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Those randomized to RIPC will undergo a standard protocol of 4 cycles of 5 minutes of forearm ischemia with 5 minutes of reperfusion requiring 35 minutes for an application. Forearm ischemia will be induced by a blood pressure cuff inflated to 200mmHg or at least 15mmHg higher than the systolic pressure if systolic > 185mmHg or until the radial pulse is obliterated. This can occur during anesthesia induction and incision/dissection prior to manipulation or clamping of the carotid.
  Arms: Remote Ischemic Preconditioning

SUMMARY:
This is a randomized controlled trial designed to test an intervention (Remote ischemic preconditioning) in patients undergoing carotid endarterectomy (CEA) for carotid artery stenosis (CAS). The outcomes of interest include neurocognitive function, cardiac complications, and biomarkers of brain ischemia.

DETAILED DESCRIPTION:
Multiple large, high quality randomized trials have shown carotid endarterectomy (CEA) is effective in decreasing future risk of stroke in patients with carotid artery stenosis. Outcomes after carotid endarterectomy have improved over time. The major risks including stroke and myocardial infarction (MI) are rare (<3% stroke and 4% for MI. However, subtle degrees of cerebral ischemia and myocardial injury are more common. Research is now focused finding ways to reduce these subclinical adverse effects of CEA.

Due to its high metabolic activity, the brain is especially vulnerable to periods of ischemia during carotid cross clamping. Ischemic tolerance has been demonstrated after direct ischemic conditioning in the brain. However, direct conditioning is difficult and potentially dangerous when is comes to carotid interventions making remote ischemic preconditioning an attractive alternative. In animal models, remote ischemic preconditioning (RIPC) has been shown to produce an equivalent response to direct neuronal conditioning at the cellular level.

The precise mechanisms underlying the phenomenon of RIPC have yet to be fully elucidated. However, It is likely that both neural and humoral mechanisms are at play. Multiple studies have shown decreased levels of inflammatory markers in brains of animal models undergoing RIPC and then middle cerebral artery occlusion.

There has only been one study of RIPC in carotid endarterectomy so far. Patients were randomized to 10 min ischemia on each leg prior to clamping the carotid. Primary outcome was significant postoperative deterioration in saccadic latency determined by quantitative oculometry (time taken to respond and fix on a visual stimulus that appears suddenly). Additionally, troponins were drawn up to 48 hours post operatively. There was deterioration in quantitative oculometry in 8/25 RIPC and 16/30 control (p=0.11) and no difference in troponins. However this was a small number of patients.

Major clinical events such as stroke or MI are uncommon following CEA. This hampers the assessment of new, novel interventions as any trial would require several thousand patients to detect a useful clinical effect. The only alternative is to use surrogate end points to obtain "proof of concept" justifying larger trials. Several serum markers of neuronal damage such as S100-beta and neuron-specific enolase have been identified but are not reliable or specific enough to be used clinically. Another surrogate that is directly related to the concept of subtle degrees of neuronal ischemia occurring during CEA is neurocognitive function.

20-25% of patients have been shown to experience significant cognitive decline following CEA. This has been correlated with findings of ischemia on diffusion weighted MRI in patients after CEA indicating that local ischemia and microemboli are responsible for this decline. Thus, neurocognitive testing before and after carotid revascularization may be an ideal surrogate end point to study in remote ischemic preconditioning and it's potential to mediate the subtle degree of neuronal ischemia produced during carotid revascularization. However, neurocognitive function is also an endpoint with clinical relevance to patients.

This study will be a double armed randomized trial. The treatment arm will be Remote ischemic preconditioning and the Control arm will be Usual care. Intervention allocation ratio will be 1:1 RIPC:usual care. Randomization strategy will be a using a 1:1 fixed block of 4 randomization stratified by symptom status and age. Those randomized to RIPC will undergo a standard protocol of 4 cycles of 5 minutes of forearm ischemia with 5 minutes of reperfusion requiring 35 minutes for an application. Forearm ischemia will be induced by a blood pressure cuff inflated to 200 millimeters of mercury (mmHg) or at least 15mmHg higher than the systolic pressure if systolic > 185mmHg or until the radial pulse is obliterated. This can occur during anesthesia induction and incision/dissection prior to manipulation or clamping of the carotid.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing carotid endarterectomy
* Indication for surgery must be symptomatic disease with >50% stenosis by duplex ultrasound or asymptomatic disease with >60% stenosis by duplex ultrasound

Exclusion Criteria:

* Lack of radial pulse on either arm
* Known Deep venous thrombosis (DVT) in arm
* Arteriovenous fistula or graft in both arms
* Diagnosed hypercoagulable state
* Pre-existing lymphedema or axillary node dissection both arms
* Diagnosis of dementia, intellectual disability, or mental illness including depression, anxiety, or schizophrenia
* Simultaneous coronary artery bypass grafting

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Immediate change in Neurocognitive function | 1 month before surgery and post operative day 1
  Montreal cognitive assessment
Longterm change in Neurocognitive function | 1 month before surgery and 1 month post operatively
  Montreal cognitive assessment

SECONDARY OUTCOMES:
S100-beta biomarker | Post operative day one
  serum level of S100-beta
Troponin | post operative day one
  serum troponin level
Stroke | within 30 days post operative
  Stroke diagnosed by MRI findings of new stroke (obtained if symptomatic)
Neuron specific enolase (NSE) biomarker | Post operative day one
  Serum level of NSE
Adverse cardiac events | 30 days postoperative
  Any new myocardial infarction, new arrhythmia, or new onset heart failure
Severity of stroke | 30 days postoperative
  National Institute of Health Stroke Scale

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Sridharan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothwell PM, Eliasziw M, Gutnikov SA, Fox AJ, Taylor DW, Mayberg MR, Warlow CP, Barnett HJ; Carotid Endarterectomy Trialists' Collaboration. Analysis of pooled data from the randomised controlled trials of endarterectomy for symptomatic carotid stenosis. Lancet. 2003 Jan 11;361(9352):107-16. doi: 10.1016/s0140-6736(03)12228-3. PMID 12531577
- [Background] LaMuraglia GM, Brewster DC, Moncure AC, Dorer DJ, Stoner MC, Trehan SK, Drummond EC, Abbott WM, Cambria RP. Carotid endarterectomy at the millennium: what interventional therapy must match. Ann Surg. 2004 Sep;240(3):535-44; discussion 544-6. doi: 10.1097/01.sla.0000137142.26925.3c. PMID 15319725
- [Background] Kragsterman B, Parsson H, Lindback J, Bergqvist D, Bjorck M; Swedish Vascular Registry (Swedvasc). Outcomes of carotid endarterectomy for asymptomatic stenosis in Sweden are improving: Results from a population-based registry. J Vasc Surg. 2006 Jul;44(1):79-85. doi: 10.1016/j.jvs.2006.03.003. Epub 2006 May 6. PMID 16682166
- [Background] Dellagrammaticas D, Lewis S, Colam B, Rothwell PM, Warlow CP, Gough MJ; GALA trial collaborators. Carotid endarterectomy in the UK: acceptable risks but unacceptable delays. Clin Med (Lond). 2007 Dec;7(6):589-92. doi: 10.7861/clinmedicine.7-6-589. PMID 18193707
- [Background] Inoue T, Ohwaki K, Tamura A, Tsutsumi K, Saito I, Saito N. Subclinical ischemia verified by somatosensory evoked potential amplitude reduction during carotid endarterectomy: negative effects on cognitive performance. J Neurosurg. 2013 May;118(5):1023-9. doi: 10.3171/2013.1.JNS121668. Epub 2013 Mar 1. PMID 23451902
- [Background] Faries PL, DeRubertis B, Trocciola S, Karwowski J, Kent KC, Chaer RA. Ischemic preconditioning during the use of the PercuSurge occlusion balloon for carotid angioplasty and stenting. Vascular. 2008 Jan-Feb;16(1):1-9. doi: 10.2310/6670.2008.00012. PMID 18258156
- [Background] Steiger HJ, Hanggi D. Ischaemic preconditioning of the brain, mechanisms and applications. Acta Neurochir (Wien). 2007 Jan;149(1):1-10. doi: 10.1007/s00701-006-1057-1. Epub 2006 Dec 14. PMID 17151832
- [Background] Vlasov TD, Korzhevskii DE, Polyakova EA. Ischemic preconditioning of the rat brain as a method of endothelial protection from ischemic/repercussion injury. Neurosci Behav Physiol. 2005 Jul;35(6):567-72. doi: 10.1007/s11055-005-0095-0. PMID 16342612
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Background] Gonzalez NR, Connolly M, Dusick JR, Bhakta H, Vespa P. Phase I clinical trial for the feasibility and safety of remote ischemic conditioning for aneurysmal subarachnoid hemorrhage. Neurosurgery. 2014 Nov;75(5):590-8; discussion 598. doi: 10.1227/NEU.0000000000000514. PMID 25072112
- [Background] Walsh SR, Tang TY, Kullar P, Jenkins DP, Dutka DP, Gaunt ME. Ischaemic preconditioning during cardiac surgery: systematic review and meta-analysis of perioperative outcomes in randomised clinical trials. Eur J Cardiothorac Surg. 2008 Nov;34(5):985-94. doi: 10.1016/j.ejcts.2008.07.062. Epub 2008 Sep 9. PMID 18783958
- [Background] Healy DA, Clarke Moloney M, McHugh SM, Grace PA, Walsh SR. Remote ischaemic preconditioning as a method for perioperative cardioprotection: concepts, applications and future directions. Int J Surg. 2014 Oct;12(10):1093-9. doi: 10.1016/j.ijsu.2014.08.352. Epub 2014 Aug 21. PMID 25152442
- [Background] Le Page S, Bejan-Angoulvant T, Angoulvant D, Prunier F. Remote ischemic conditioning and cardioprotection: a systematic review and meta-analysis of randomized clinical trials. Basic Res Cardiol. 2015 Mar;110(2):11. doi: 10.1007/s00395-015-0467-8. Epub 2015 Feb 5. PMID 25653117
- [Background] Walsh SR, Nouraei SA, Tang TY, Sadat U, Carpenter RH, Gaunt ME. Remote ischemic preconditioning for cerebral and cardiac protection during carotid endarterectomy: results from a pilot randomized clinical trial. Vasc Endovascular Surg. 2010 Aug;44(6):434-9. doi: 10.1177/1538574410369709. Epub 2010 May 18. PMID 20484064
- [Background] Sahlein DH, Heyer EJ, Rampersad A, Winfree CJ, Solomon RA, Benvenisty AI, Quest DO, Du E, Connolly ES. Failure of intraoperative jugular bulb S-100B and neuron-specific enolase sampling to predict cognitive injury after carotid endarterectomy. Neurosurgery. 2003 Dec;53(6):1243-9 discussion 1249-50. doi: 10.1227/01.neu.0000093493.16850.11. PMID 14633290
- [Background] Connolly ES Jr, Winfree CJ, Rampersad A, Sharma R, Mack WJ, Mocco J, Solomon RA, Todd G, Quest DO, Stern Y, Heyer EJ. Serum S100B protein levels are correlated with subclinical neurocognitive declines after carotid endarterectomy. Neurosurgery. 2001 Nov;49(5):1076-82; discussion 1082-3. doi: 10.1097/00006123-200111000-00010. PMID 11846900
- [Background] Rasmussen LS, Christiansen M, Johnsen J, Gronholdt ML, Moller JT. Subtle brain damage cannot be detected by measuring neuron-specific enolase and S-100beta protein after carotid endarterectomy. J Cardiothorac Vasc Anesth. 2000 Apr;14(2):166-70. doi: 10.1016/s1053-0770(00)90012-0. PMID 10794336
- [Background] Missler U, Wiesmann M, Friedrich C, Kaps M. S-100 protein and neuron-specific enolase concentrations in blood as indicators of infarction volume and prognosis in acute ischemic stroke. Stroke. 1997 Oct;28(10):1956-60. doi: 10.1161/01.str.28.10.1956. PMID 9341703
- [Background] Heyer EJ, Sharma R, Rampersad A, Winfree CJ, Mack WJ, Solomon RA, Todd GJ, McCormick PC, McMurtry JG, Quest DO, Stern Y, Lazar RM, Connolly ES. A controlled prospective study of neuropsychological dysfunction following carotid endarterectomy. Arch Neurol. 2002 Feb;59(2):217-22. doi: 10.1001/archneur.59.2.217. PMID 11843692
- [Background] Mocco J, Wilson DA, Komotar RJ, Zurica J, Mack WJ, Halazun HJ, Hatami R, Sciacca RR, Connolly ES Jr, Heyer EJ. Predictors of neurocognitive decline after carotid endarterectomy. Neurosurgery. 2006 May;58(5):844-50; discussion 844-50. doi: 10.1227/01.NEU.0000209638.62401.7E. PMID 16639318
- [Background] Baracchini C, Mazzalai F, Gruppo M, Lorenzetti R, Ermani M, Ballotta E. Carotid endarterectomy protects elderly patients from cognitive decline: a prospective study. Surgery. 2012 Jan;151(1):99-106. doi: 10.1016/j.surg.2011.06.031. Epub 2011 Sep 22. PMID 21943640
- [Background] Qu L, Feng J, Zou S, Bai J, Hu Z, Guo M, Jing Z. Improved visual, acoustic, and neurocognitive functions after carotid endarterectomy in patients with minor stroke from severe carotid stenosis. J Vasc Surg. 2015 Sep;62(3):635-44.e2. doi: 10.1016/j.jvs.2015.04.401. Epub 2015 Jun 10. PMID 26070604
- [Background] Wilson DA, Mocco J, D'Ambrosio AL, Komotar RJ, Zurica J, Kellner CP, Hahn DK, Connolly ES, Liu X, Imielinska C, Heyer EJ. Post-carotid endarterectomy neurocognitive decline is associated with cerebral blood flow asymmetry on post-operative magnetic resonance perfusion brain scans. Neurol Res. 2008 Apr;30(3):302-6. doi: 10.1179/016164107X230540. Epub 2007 Sep 4. PMID 17803842
- [Background] De Rango P, Caso V, Leys D, Paciaroni M, Lenti M, Cao P. The role of carotid artery stenting and carotid endarterectomy in cognitive performance: a systematic review. Stroke. 2008 Nov;39(11):3116-27. doi: 10.1161/STROKEAHA.108.518357. Epub 2008 Aug 21. PMID 18723423
- [Background] Paraskevas KI, Lazaridis C, Andrews CM, Veith FJ, Giannoukas AD. Comparison of cognitive function after carotid artery stenting versus carotid endarterectomy. Eur J Vasc Endovasc Surg. 2014 Mar;47(3):221-31. doi: 10.1016/j.ejvs.2013.11.006. Epub 2013 Nov 28. PMID 24393665
- [Background] Wang Q, Zhou M, Zhou Y, Ji J, Raithel D, Qiao T. Effects of Carotid Endarterectomy on Cerebral Reperfusion and Cognitive Function in Patients with High Grade Carotid Stenosis: A Perfusion Weighted Magnetic Resonance Imaging Study. Eur J Vasc Endovasc Surg. 2015 Jul;50(1):5-12. doi: 10.1016/j.ejvs.2015.03.032. Epub 2015 Apr 29. PMID 25933475